CLINICAL TRIAL: NCT04075435
Title: Open-Label Trial of a Cannabidiol Solution for the Treatment of Behavioral Symptoms in Older Adults With Mild Cognitive Impairment or Alzheimer's Dementia
Brief Title: Cannabidiol Solution for the Treatment of Behavioral Symptoms in Older Adults With Mild Cognitive Impairment or Alzheimer's Dementia
Acronym: CBD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Spier Family Foundation (Unknown)
Responsible Party: Principal Investigator, Staci Gruber, Ph.D., Directory, Cognitive and Clinical Neuroimaging Core; Director, Marijuana Investigations for Neuroscientific Discovery (MIND), Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P002466
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Anxiety; Agitation,Psychomotor; Mild Cognitive Impairment (MCI) Due to Alzheimer's Disease
Keywords: cannabidiol; older adults; dementia
MeSH Terms: conditions — Alzheimer Disease; Anxiety Disorders; Psychomotor Agitation; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: This is an open label trial; all participants will receive active drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All subjects (Other): This arm will include all subjects, individuals will administer a high CBD, low THC full spectrum sublingual solution twice daily on a variable dosing schedule.
  Interventions: Drug: high CBD/low THC sublingual solution

INTERVENTIONS:
Drug: high CBD/low THC sublingual solution — Hemp derived solution to be administered sublingually twice daily.

SUMMARY:
This is an open label, eight week, clinical trial of a proprietary high CBD/low THC sublingual solution for the treatment of clinically significant anxiety and agitation in individuals with mild cognitive impairment (MCI) or mild to moderate Alzheimer's Disease (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of probable Alzheimer's Dementia via criteria from McKhann et al., or MCI
2. MMSE score of 15-30 (inclusive)
3. Clinically significant degree of anxiety, as defined by a Clinical Impression total column score of ≥4 on the Anxiety domain of the NPI-C
4. A health care proxy available to sign consent on behalf of the participant (if applicable)
5. A caregiver who spends at least 10 hours per week with the subject who is able to attend all study visits
6. Participants and their study partner must be fluent in English
7. Must be 55-90 years old (inclusive)

Exclusion Criteria:

1. Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease, which might confound assessment of safety outcomes.
2. Seizure disorder
3. Lifetime diagnosis of bipolar disorder, schizophrenia, schizoaffective disorder, as determined by the MINI
4. Current episode of major depression, as determined by the MINI
5. Active substance abuse or dependence within the past 6 months, as determined by the MINI
6. Delirium (as measured by the CAM)
7. Current inpatient hospitalization
8. Current regular use of cannabinoid products (>1 use per month)
9. Positive urine screen for THC at the screening or baseline visit
10. Allergy to coconut
11. Participants taking strong inhibitors or inducers of CYP3A4 (e.g. fluconazole, fluoxetine, fluvoxamine, ticlopidine, St. John's Wort, etc.), CYP2C19 (ketoconazole, erythromycin, etc.), or anti-epileptic drugs

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2026-01-16 (Estimated); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
Total of clinician impression column on anxiety domain of the NPI-C | Continuous, weeks 0-8
  Measure of Anxiety Domain on the Neuropsychiatric Inventory-Clinician scale

SECONDARY OUTCOMES:
Total score on the Generalized Anxiety Disorder 7 scale | Continuous, week 0-8
  Secondary Outcome Measure of anxiety reduction
Number of serious adverse events | Continuous, weeks 0-8
  Secondary Outcome Measure of safety defined by absence of serious adverse events
Week 8 MMSE total score compared to baseline MMSE total score | longitudinal: screening/baseline and week8
  Secondary Outcome Measure of safety as defined by lack of treatment emergent cognitive impairment as measured by the Mini Mental Status Exam (MMSE)
Score on the confusion assessment method | Continuous screening weeks 0-8, dichotomous
  Secondary Outcome Measure of safety defined as absence of treatment emergent delirium as measured by the Confusion Assessment Method (CAM)
Number and severity of side effects reported | Continuous, weeks 0-8
  Secondary Outcome Measure of safety defined as a low number of emergent somatic side effects as measured by the Medication Side Effects Questionnaire

OTHER OUTCOMES:
Total clinical impression column score on neuropsychiatric inventory agitation and aggression domains (NPI-C) | Continuous, weeks 0-8
  Exploratory measure to see reduction in agitation and aggression symptoms
Total score of Cohen-Mansfield Inventory (CMAI) | Continuous, weeks 0-8
  Exploratory measure to see reduction in agitation symptoms
Total Score of Zarit Caregiver Burden Interview | Continuous, weeks 0-8
  Exploratory downstream reduction in caregiver burden
Stability of anxiety and agitation reduction using anxiety domain of NPI-C and GAD-7 | Months 3, 6, 9, and 12 of the optional follow-up phase
  Exploratory investigation into the stability of anxiety reduction using the anxiety domain score on the NPI-C and the GAD-7 during the optional follow-up phase
Stability of caregiver burden reduction | Months 3, 6, 9, and 12 of the optional follow-up phase
  Exploratory investigation into reduction of caregiver burden using the Zarit Caregiver Burden Interview during the optional follow-up phase

CONTACTS AND LOCATIONS:
Overall Officials: Staci Gruber, PhD, Principal Investigator — Mclean Hospital; Ipsit V Vahia, MD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No